CLINICAL TRIAL: NCT03604146
Title: Establishment of Quality Control Index System and Strategy for Chronic Obstructive Pulmonary Disease in China
Brief Title: Quality Control for Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Fengyan Wang, Principal Investigator, Guangzhou Institute of Respiratory Disease
Other Study IDs: C2017050
Record Dates: First submitted 2018-07-10; First posted 2018-07-27 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: COPD
Keywords: COPD; Quality Control
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: Doctors and nurses were trained to treat chronic obstructive pulmonary disease according to the GOLD guidelines.Hospital patient cohort and outpatient cohort will be setted. Subjects were interviewed and received pulmonary function tests.
- Intervention group: Doctors and nurses will not receive any training from research team. Hospital patient cohort and outpatient cohort will be setted. Subjects were interviewed and received pulmonary function tests.
  Interventions: Behavioral: Medical quality control intervention strategy

INTERVENTIONS:
Behavioral: Medical quality control intervention strategy — Training and education for diagnosis, treatment and management of COPD for doctors and nurses; Regular inspection and supervision of medical quality
  Groups: Intervention group

SUMMARY:
This is a 1 year longitudinal study to establish a related index system for chronic obstructive pulmonary disease(COPD) quality control.Clinical and economic data of COPD patients will be collected and analyzed.

DETAILED DESCRIPTION:
Sixteen hospitals in Guangdong Province were randomly divided into control group and intervention group.Doctors and nurses of intervention group were trained treat chronic obstructive pulmonary disease according to the GOLD(Global InitiaTive of Chronic Obstructive Lung Disease) guidelines，while those in the control group will not receive any training from research team. Hospital patient cohort and outpatient cohort will be setted. Subjects were interviewed and received pulmonary function tests.All patients will be followed and events of acute exacerbation will be recorded.Factors that influence patient prognosis and economic-health benefits will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients was diagnosed as COPD according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines older than 40 years old.Patients was hospitalized for AECOPD or visiting outpatient department for COPD.

  * A signed and dated written informed consent is obtained prior to participation.
  * Able to comply with the requirements of the protocol and be available for study visits over 1 years.

Exclusion Criteria:

A COPD subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Known respiratory disorders, or disorders identified at screening/visit

  1 (including identification on the first CT scan), other than COPD (e.g.: lung cancer, sarcoidosis, tuberculosis, lung fibrosis, cystic fibrosis)
* Having undergone lung surgery (e.g. lung reduction, lung transplant)
* Severe liver and kidney dysfunction
* Have cancer or have had cancer in the 5 years prior to study entry
* Taking part in a blinded drug study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Grade II - III hospital in Guangdong Province
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
rate of exacerbations of COPD (AECOPD) | 1 year
  The rate of exacerbations within 1 year in the intervention group and the control group will be tracked.

SECONDARY OUTCOMES:
rate of readmission for AECOPD | 1 year
  The rate of readmission for AECOPD within 1 year in the intervention group and the control group will be tracked.
change of Forced expiratory volume in one second(FEV1) | 1 year
  The difference in FEV1 after bronchodilator between baseline and 1 year later

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, MD, Study Director — Guangzhou Institute of Respiratory Health,The First Affiliated Hospital of Guangzhou Medical University,China
Locations (1):
- Guangzhou Institute of Respiratory Health,The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China